CLINICAL TRIAL: NCT01766440
Title: Pharmacokinetics and Pharmacodynamics of Calcitriol 3 mcg/g Ointment Applied Twice Daily for 14 Days Under Conditions of Maximal Use in Pediatric Subjects (2 to 12 Years of Age) With Plaque Psoriasis
Brief Title: PK and PD Study of Calcitriol 3 mcg/g Ointment in Pediatric Subjects With Plaque Psoriasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RD.06. SPR.18104
Record Dates: First submitted 2013-01-09; First posted 2013-01-11 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2017-04

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Calcitriol; Ointments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcitriol 3 mcg/g ointment (Experimental): Topical application every 12 hours for 14 consecutive days
  Interventions: Drug: Calcitriol 3 mcg/g ointment

INTERVENTIONS:
Drug: Calcitriol 3 mcg/g ointment — Topical ointment; twice daily application

SUMMARY:
The purpose of this study is to determine if the calcitriol absorption in pediatric subjects is comparable to that in adults and adolescents, with no significant impact on calcium/phosphorus metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pediatric subjects, 2 to 12 years of age inclusive at screening
* Clinical diagnosis of plaque type psoriasis involving 3% through 35% body surface area at screening and baseline (excluding face and scalp)

Exclusion Criteria:

* Subjects with guttate or pustular psoriasis, erythrodermic psoriasis or active infection
* Vitamin D deficiency at screening
* Subjects with hypercalcemia and out of range urinary calcium/creatinine ratio at screening
* Subjects with secondary hyperparathyroidism at screening

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, M.D., Study Director — Galderma R&D, LLC
Locations (8):
- United States (8):
  - Rady Children's Hospital - Pediatric and Adolescent Dermatology, San Diego, California
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - University of North Carolina Dermatology and Skin Cancer Center, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Menter Dermatology Research Institute, Dallas, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calcitriol 3 mcg/g Ointment
Started | 18
Completed | 17
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Calcitriol 3 mcg/g Ointment
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.4 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Calcitriol Plasma Level
Description: Cmax of calcitriol plasma level at Day 14 (Peak plasma concentration of calcitriol from Day 1 to Day 14)
Time Frame: Day 14
Population: Safety population: All enrolled subjects having received the treatment at least once.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Calcitriol 3 mcg/g Ointment
Number analyzed (Participants) | 17
pg/mL | 120.7 (31.5)

2. Primary Outcome: Cmin of Calcitriol Plasma Level
Description: Cmin of calcitriol plasma level at Day 14
Time Frame: Day 14
Population: Safety population: All enrolled subjects having received the treatment at least once.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Calcitriol 3 mcg/g Ointment
Number analyzed (Participants) | 17
pg/mL | 92.6 (24.2)

3. Primary Outcome: Tmax of Calcitriol Plasma Level
Description: Tmax of calcitriol plasma level at Day 14
Time Frame: Day 14
Population: Safety population: All enrolled subjects having received the treatment at least once.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Calcitriol 3 mcg/g Ointment
Number analyzed (Participants) | 17
hour | 1.46 (2.36)

4. Primary Outcome: AUC (0-6h) of Calcitriol Plasma Level
Description: AUC (0-6h) of calcitriol plasma level at Day 14 (Pre-dose to 6 hours post-dose)
Time Frame: Day 14
Population: Safety population: All enrolled subjects having received the treatment at least once.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Calcitriol 3 mcg/g Ointment
Number analyzed (Participants) | 17
pg*h/mL | 650.3 (166.8)

5. Primary Outcome: AUC (0-9h) of Calcitriol Plasma Level
Description: AUC (0-9h) of calcitriol plasma level at Day 14 (Pre-dose to 9 hours post-dose. For subjects with a body weight of <15 kg, AUC (0-9h) was extrapolated based on the pre-dose to 6 hours post-dose PK samples.)
Time Frame: Day 14
Population: Safety population: All enrolled subjects having received the treatment at least once.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Calcitriol 3 mcg/g Ointment
Number analyzed (Participants) | 17
pg*h/mL | 952.6 (235.9)

6. Primary Outcome: AUC (0-12h) of Calcitriol Plasma Level
Description: AUC (0-12h) of calcitriol plasma level at Day 14 (For subjects with a body weight of < 15 kg, AUC (0-9h) was extrapolated based on the pre-dose to 6 hours post dose PK samples. For subjects with a body weight of ≥ 15 kg, AUC (0-12h) was extrapolated based on the pre-dose to 9 hours post-dose PK samples.)
Time Frame: Day 14
Population: Safety population: All enrolled subjects having received the treatment at least once.
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Calcitriol 3 mcg/g Ointment
Number analyzed (Participants) | 17
pg*h/mL | 1268.9 (307.3)

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Calcitriol 3 mcg/g Ointment
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 9/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcitriol 3 mcg/g Ointment (N=18)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated early due to slow enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No